CLINICAL TRIAL: NCT06630416
Title: A Phase II Trial to Evaluate Pemetrexed Response in Relation to Tumor Alterations of Gene Status in Patients With Previously Treated Metastatic Urothelial Carcinoma and Other Solid Tumors
Brief Title: Pemetrexed Response in Relation to Tumor Alterations of Gene Status for the Treatment of Patients With Metastatic Urothelial Bladder Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 24MH03; NCI-2024-07862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00222531; NU 24MH03 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Bladder Urothelial Carcinoma; Metastatic Malignant Solid Neoplasm; Stage IV Bladder Cancer AJCC v8
MeSH Terms: conditions — Neoplasm Metastasis; Urinary Bladder Neoplasms | interventions — Specimen Handling; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pemetrexed) (Experimental): Patients receive pemetrexed IV over 10 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and urine sample collection on study as well as CT throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Pemetrexed

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy

SUMMARY:
This phase II trial tests how well pemetrexed works in treating patients with urothelial bladder cancer and other solid tumors that have spread from where they first started (primary site) to other places in the body (metastatic) with mutations that result in a loss of function in the MLL4-protein/KMT2D-gene or UTX-protein/KDM6A-gene or MTAP enzyme. Loss of function due to a genetic mutation means a gene's activity may be reduced or eliminated. Mutations that result in a loss of function in the MLL4-protein or KMT2D-gene are found in 9.96% of all cancers including bladder carcinoma patients, esophageal squamous cell carcinoma and esophageal adenocarcinoma patients. In addition, mutations that result in a loss of function in the UTX-protein or KDM6A-gene are found in approximately 5% of all tumors, including bladder cancers, endometrial cancer, and esophagogastric cancer amongst many other tumor types. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by stopping cells from using folic acid to make deoxyribonucleic acid and may kill tumor cells. Giving pemetrexed may increase response in patients with metastatic urothelial bladder cancer and other solid tumors with the loss of function in the MLL4-protein/KMT2D-gene or UTX-protein/KDM6A-gene or MTAP enzyme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) in patients with metastatic solid tumors and MLL4-protein (KMT2D-gene) and UTX-protein (KDM6A-gene) or MTAP loss of function mutations treated with pemetrexed will assess pemetrexed.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) for patients with metastatic solid tumors and MLL4-protein (KMT2D-gene) and UTX-protein (KDM6A-gene) or MTAP loss of function mutations treated with pemetrexed.

II. To determine the overall survival (OS) for patients with metastatic solid tumors and MLL4-protein (KMT2D-gene) and UTX-protein (KDM6A-gene) or MTAP loss of function mutations treated with pemetrexed.

III. To determine the duration of response (DOR) for patients with metastatic solid tumors and MLL4-protein (KMT2D-gene) and UTX-protein (KDM6A-gene) or MTAP loss of function mutations treated with pemetrexed.

IV. To assess safety and tolerability of pemetrexed in patients with metastatic solid treated with pemetrexed.

EXPLORATORY OBJECTIVE:

I. To collect plasma and urine samples for future translational studies to determine mechanisms of resistance to pemetrexed.

OUTLINE:

Patients receive pemetrexed intravenously (IV) over 10 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood and urine sample collection on study as well as computed tomography (CT) throughout the trial.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically or cytologically confirmed metastatic urothelial bladder carcinoma (Arm A) or other metastatic solid malignancy (Arm B) and MLL4-protein (KMT2D-gene) and UTX-protein (KDM6A-gene) or MTAP loss of function mutation including but not limited to single nucleotide variant (SNVs) that cause truncation, copy number variations (CNVs), and indels confirmed by next generation sequencing or immunohistochemistry techniques
* Patients must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), measured preferably by computed tomography (CT) scan
* Patients who have received any prior neoadjuvant or systemic chemotherapy are eligible.

  * Notes:

    * Patients must have progressive disease despite two prior lines of therapy in the metastatic setting unless the patient was not suitable for an approved second line regimen due to intolerance or another clinical factor;
    * Treatment cannot have included prior pemetrexed. Any prior intravesical therapy, or immunotherapy is allowed. At least 4 weeks (28 days) wash-out period since prior chemotherapy or radiation therapy or targeted agent is required
* Patients must be aged ≥ 18 years
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (growth factor allowed and can be added at the discretion of the treating oncologist)
* Hemoglobin (Hgb) ≥ 8.5 g/dL (without the need for transfusion within the previous one week)
* Platelets (PLT) ≥ 100,000/mL (without the need for platelet transfusion within the previous one week)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), except subjects with Gilbert's syndrome or liver metastases, who must have a baseline total bilirubin ≤ 3.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 3 x institutional ULN or ≤ 5 x ULN if documented liver metastases are present
* Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN or ≤ 5 x ULN if documented liver metastases are present
* Creatinine clearance ≥ 45 mL/min/1.73 m^2 using the standard Cockcroft and Gault formula
* Patients must have the ability to comply with the administration of supplemental therapies including folic acid, vitamin B12 and steroids as directed by study team and as per standard of care and institutional standards and practice for pemetrexed use
* Patients must be able swallow oral medication or not have problems/diseases that affect absorption or oral medication
* Patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration. Please note this lab is not a requirement for eligibility, however, if it was previously done as part of the patient's health care, it should be documented for eligibility
* Patients with a known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Please note this lab is not a requirement for eligibility, however, if the lab has been completed previously as part of the patient's health care, then it should be documented for eligibility
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with a known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. Please note this lab is not a requirement for eligibility, however if it was previously done as part of the patient's health care, it should be documented for eligibility
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Pemetrexed is known to be teratogenic. For this reason, patients of child-bearing potential (POCBP) and their partners with sperm-producing reproductive capacity must agree to use adequate contraception from time of informed consent, for the duration of study participation, and for 180 days following completion of pemetrexed therapy. Should a POCBP become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately. Patients with sperm-producing reproductive capacity (PWSPRC) treated or enrolled on this protocol must also agree to use adequate contraception with partners of childbearing potential from time of informed consent, for the duration of study participation, and 180 days after completion of administration

  * Note: A POCBP is any patient (regardless of gender, sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) with an egg-producing reproductive tract who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative pregnancy test prior to registration on study
* The ability to interrupt nonsteroidal anti-inflammatory drugs (NSAIDS) or aspirin at higher dose (> 1.3 g per day) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed
* Patients must be able to understand and voluntarily sign a written informed consent and willing and able to comply with the protocol requirements including scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Patients who received prior pemetrexed containing chemotherapy
* Patients who have had chemotherapy or radiotherapy ≤ 28 days (prior to planned treatment start date)
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia, neuropathy and other non-significant adverse events deemed not clinically significant by the treating investigator, adverse events per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v 5.0)
* Patients who are receiving any other investigational agents. A 28 day wash out period will be required after discontinuation of an investigational agent prior to first day of study treatment
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pemetrexed
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification

  * Note: To be eligible for this trial, patients should be class 2B or better
* Patients with presence of third space fluid which cannot be controlled by drainage

  * Note: For patients who develop or have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before or during initiation of pemetrexed therapy, consideration should be given to draining the effusion prior to dosing. However, if, in the investigator's opinion, the effusion represents progression of disease, the patient should be discontinued from study therapy
* Has received the final dose of any of the following treatments/ procedures with the specified minimum intervals before first dose of study drug:

  * Focal radiation therapy - 7 days
  * Surgery with general anesthesia - 7 days
  * Surgery with local anesthesia - 3 days
* Patients of child bearing (POCB) potential who are pregnant or nursing.

  * Note: Registration of patients is completed in Northwestern Oncology Trial Information System (NOTIS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2029-05-10 (Estimated); Study Completion 2030-05-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From baseline until the subject experiences disease progression, the subject initiates subsequent anti-cancer therapy, or the subject completes study participation (whichever occurs first), assessed up to 12 months
  ORR is defined as the proportion of treated patients who experience an objective response (complete response [CR] or partial response [PR]). The date of first response for either CR or PR will be used to calculate ORR. Will be measured every 9 weeks +/- 10 days according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). CR and PR need to be confirmed by a subsequent scan. Will compute two-sided 90% confidence intervals (CIs) for ORR using the exact binomial method. The statistical significance of the ORR will be assessed using chi-square tests or Fisher's exact tests, depending on the sample size.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from the start of treatment to the first documented progression or death from any cause, whichever comes first, assessed up to 12 months
  PFS will be analyzed using Kaplan-Meier survival analysis to estimate the survival distribution. The median PFS and corresponding 95% confidence intervals will be reported. Log-rank tests will be used to compare PFS between different subgroups. Additionally, Cox proportional hazards models will be used to evaluate the impact of various covariates on PFS, providing hazard ratios (HRs) and 95% CIs.
Overall survival (OS) | Time from the start of treatment to death from any cause, assessed up to 12 months
  OS will be analyzed using Kaplan-Meier survival analysis. The median OS and corresponding 95% confidence intervals will be reported. Log-rank tests will be utilized to compare OS between different subgroups. Cox proportional hazards models will also be employed to assess the effect of covariates on OS, with results presented as HRs and 95% CIs.
Duration of response (DOR) | Time from first response (complete or partial) until progression or death, assessed up to 12 months
  DOR will be assessed by disease progression, defined as experiencing progressive disease per RECIST v1.1, or death due to disease. If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy the DOR will be censored as the last available disease assessment based on clinical or radiographic evaluation.
Incidence of adverse events | Up to 12 months
  Will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and will be documented by clinical or radiographic evaluation or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States